CLINICAL TRIAL: NCT02700347
Title: Evaluating Pharmacokinetics and Whole Blood Bactericidal Activity Against Mycobacterium Tuberculosis of Pyrazinamide Boosted With Allopurinol in Healthy Volunteers
Brief Title: Whole Blood Bactericidal Activity Against Mycobacterium Tuberculosis of Pyrazinamide Plus Allopurinol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PZA_WBA
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Pyrazinamide; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose pyrazinamide (Experimental): Day 0: Pyrazinamide 10mg/kg, Day 5: Allopurinol 100mg single dose, Day 6: Allopurinol 100mg single dose, Day 7: Pyrazinamide 10mg/kg plus allopurinol 100mg single dose, Day 8: Allopurinol 100mg single dose.
  Interventions: Drug: Pyrazinamide; Drug: Allopurinol
- Standard dose pyrazinamide (Experimental): Day 0: Pyrazinamide 25mg/kg single dose, Day 5: Allopurinol 100mg single dose, Day 6: Allopurinol 100mg single dose, Day 7: Pyrazinamide 25mg/kg plus allopurinol 100mg single dose, Day 8: Allopurinol 100mg single dose.
  Interventions: Drug: Pyrazinamide; Drug: Allopurinol
- High dose pyrazinamide (Experimental): Day 0: Pyrazinamide 35mg/kg single dose, Day 5: Allopurinol 100mg single dose, Day 6: Allopurinol 100mg single dose, Day 7: Pyrazinamide 35mg/kg plus allopurinol 100mg single dose, Day 8: Allopurinol 100mg single dose.
  Interventions: Drug: Pyrazinamide; Drug: Allopurinol

INTERVENTIONS:
Drug: Pyrazinamide
Drug: Allopurinol

SUMMARY:
The purpose of this study is to evaluate the bactericidal activity against Mycobacterium tuberculosis of pyrazinamide in combination with allopurinol. Pharmacokinetics (PK) and whole blood bactericidal activity (WBA) will be measured in healthy volunteers following administration of pyrazinamide alone and in combination with allopurinol.

DETAILED DESCRIPTION:
The whole blood bactericidal activity (WBA) assay is an ex vivo model for measuring the combined effects of administered drugs, host factors and strain factors on mycobacterial sterilisation. If performed in parallel with PK measurements, the method can be used to evaluate the effect of drugs throughout the dosing cycle. The aim of this trial is to assess the WBA activity and PK data of pyrazinamide and its metabolites boosted with allopurinol in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 21 and 70 years old
2. Male or female willing to comply with the study visits and procedures
3. Willing and able to provide written informed consent

Exclusion Criteria:

1. Women who are currently pregnant or breastfeeding
2. Body weight 50kg or below
3. HLA-B*5801 allele positive
4. Clinical evidence (symptoms and/or signs) suggestive of active TB
5. Previous hypersensitivity, intolerance or allergy to pyrazinamide or allopurinol
6. Current use of any drugs or medication known to have an interaction with pyrazinamide or allopurinol, or known to have anti-TB activity
7. Evidence of renal or hepatic dysfunction or any clinically significant deviation from normal during screening including laboratory determinations
8. Known hepatic disease (including chronic hepatitis), recent hepatitis (within last 6 months) or alcohol abuse
9. Known hyperuricaemia or evidence of hyperuricaemia at screening
10. History or current episode of gout
11. Any other significant condition that would, in the opinion of the investigator, compromise the volunteer's safety or outcome in the trial
12. Current participation in other clinical intervention trial or research protocol

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Cumulative whole blood bactericidal activity (WBA) | 48 hours
  Cumulative bactericidal activity calculated as log change CFU.day

SECONDARY OUTCOMES:
Plasma concentrations of study drugs to determine the Area Under the Curve (AUC) | 48 hours
Plasma concentrations of study drugs to determine the Maximum Plasma Concentration (Cmax) | 48 hours
Plasma concentrations of study drugs to determine the drug half-life (t1/2) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Naftalin CM, Verma R, Gurumurthy M, Lu Q, Zimmerman M, Yeo BCM, Tan KH, Lin W, Yu B, Dartois V, Paton NI. Coadministration of Allopurinol To Increase Antimycobacterial Efficacy of Pyrazinamide as Evaluated in a Whole-Blood Bactericidal Activity Model. Antimicrob Agents Chemother. 2017 Sep 22;61(10):e00482-17. doi: 10.1128/AAC.00482-17. Print 2017 Oct. PMID 28739782